CLINICAL TRIAL: NCT01082796
Title: Investigate the Relationship Between CYP2C19 Genetic Polymorphisms and Pharmacokinetics of Glipizide in Healthy Chinese Subjects
Brief Title: Cytochrome P450 2C19 Variant is Related to Pharmacokinetics of Glipizide Extended Release Tablet in Chinese Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Academy of Sciences (Other Government)
Collaborators: LanZhou University (Other)
Responsible Party: Shanghai Institute of Materia Medica, Chinese Academy of Sciences, The First Affiliated Hospital of Lanzhou University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SIMM-DMPK-090903
Record Dates: First submitted 2010-03-04; First posted 2010-03-09 (Estimated); Last update posted 2010-03-09 (Estimated); Status verified 2009-11

CONDITIONS: Genotype; Pharmacokinetic
MeSH Terms: interventions — Glipizide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CYP2C19 EMs group (Other): cyp2c19*1/*1 carriers
  Interventions: Drug: Glipizide
- CYP2C19 PMs group (Other): cyp2c19*2/*2 or *2/*3
  Interventions: Drug: Glipizide

INTERVENTIONS:
Drug: Glipizide — Each subject received 5 mg glipizide extended release tablet once daily for 7 days.
  Other Names: Glucotrol XL®

SUMMARY:
Diabetes mellitus is a growing global disease now and future, and in China, 1.2 million peoples per year have been diagnosed as diabetes mellitus. 90% diabetes mellitus patient is Type 2 diabetes mellitus. Glipizide is a potent drug to service patients who suffer from Type 2 disease. Little information has been presented for the relationship between CYP2C19 genetic polymorphism and glipizide, since recently the investigators reported that there existed a tendency. In this study the investigators found that CYP2C19 polymorphism significantly influenced the pharmacokinetics of glipizide.

DETAILED DESCRIPTION:
Blood samples were obtained from 127 unrelated healthy male Chinese subjects in Gansu Province. After genotyping, 14 subjects (age, 19-26; weight, 59.5-70.0 kg) were enrolled in the study. They were divided into two groups, EMs homo and PMs group. There were no significant differences in age or body weight seen in the two groups.

Each subject received 5 mg glipizide extended release tablet once daily for 7 days. For the first 6 days, glipizide was administered just after a standard breakfast. On day 7, after an overnight fast, each subject received a glipizide extended released tablet (Glucotrol XL, Pfizer, USA) with 100 mL water. Standard meals were given in 4 h and 10 h after dosing. Venous blood samples were collected immediately before and at 2, 4, 6, 8, 10, 12, 14, 16, 20, 24, 36, and 48 h after dosing. Blood samples, collected in EDTA tubes, were centrifuged (2500 g) immediately for 10 min and plasma samples separated were stored at -80ºC until assay.

For safety, blood glucose levels were determined directly by use of a Glucose Meter (Accu-Chek, Roche, Germany) at 0, 2, 4, 6, 8, 10, 12, 14, 16, 20and 24 h after last dosing (on day 7).

ELIGIBILITY:
Inclusion Criteria:

* male
* healthy
* nonsmokers

Exclusion Criteria:

* BMI > 24 or BMI < 19
* had any family history of diabetes mellitus

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2009-11; Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Da F Zhong, PH.D, Study Director — Shanghai Institute of Materia Medica, Chinese Academy of Sciences
Locations (1):
- Departmant of Clinical Pharmacology, the First Affiliated Hospital of Lanzhou University, Lanzhou, Gansu, China

REFERENCES:
- See also: Our organization — http://english.simm.cas.cn/